CLINICAL TRIAL: NCT06454812
Title: The Effect of Mechanical Vibration and Helfer Skin Tap Technique on Procedural Pain in Healthy Infants During Intramuscular Vaccination: a Randomized Controlled Study
Brief Title: The Effect of Mechanical Vibration and Helfer Skin Tap Technique on Procedural Pain in Infants During Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20.09.2023/174
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Procedural Pain; Nursing Caries; Pain, Acute
Keywords: Healthy infant; Nonpharmacological pain management; Procedural pain
MeSH Terms: conditions — Pain, Procedural; Acute Pain

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to experimental and control groups using block randomization method. Body weight and sex variables will be used for block randomization.
Who Masked: Participant, Outcomes Assessor
Masking Description: Using the block randomization technique, participants will be divided into 3 groups. A web-based randomization list creation tool will be used to create the blocked randomization list. Control and intervention groups will be coded as A, B and C using the sealed envelope method. Randomization information will be kept from the researcher involved in data collection until data collection begins. The researcher will learn which group each baby is in just before the application (researcher blinding).
  Parents will know which group the baby is in within the scope of the research. By the nature of the sample group, babies are blind.
  Research data will be entered into the computer database by coding the group name as A, B and C, and statistical analysis will be performed using this coding (statistician blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): The control group will receive routine vaccinations.
- Mechanical vibration (Experimental): Mechanical vibration will be used during routine vaccination of infants in this group.
  Interventions: Device: Mechanical vibration
- Helfer skin tap technique (Experimental): Helfer skin tap technique will be used during routine vaccinations of infants in this group.
  Interventions: Behavioral: Helfer skin tap technique (HSTT)

INTERVENTIONS:
Device: Mechanical vibration — The vibration device will be placed on the procedure site (on the vastus lateralis muscle) on the left extremity and fixed through a long gauze. The vibration device will be operated for 30 seconds with reference to previous studies, then the nurse will administer routine intramuscular Hepatitis B vaccine. A gap of approximately 1-2 cm will be left between the device and the injection site. After the vaccination procedure is completed, the vibration will be terminated. The same procedure was repeated for DTaP-IPV-Hib vaccine administered to the the right extremity. The baby will be swaddled and placed in the mother's lap.
  Arms: Mechanical vibration
Behavioral: Helfer skin tap technique (HSTT) — In this group, HSTT consisting of 4-stage strokes will be applied to the vaccination site. The nurse will make approximately 10 strokes for 5 seconds with the palmar side of the fingers of the dominant hand to the injection site to relax the muscles (Stage 1). The nurse will give a V-shaped position to the thumb and index finger of the non-dominant hand and give 3 strokes to the injection site with the palmar side of the fingers (Stage 2). The skin entry site of the needle will remain inside the V-shape. Simultaneously with the 3rd stroke, the nurse will insert the needle into the muscle at a 90 degree angle. The nurse will inject the vaccine into the muscle while continuing to tap the skin with the palmar side of the fingers of the non-dominant hand (Stage 3). The nurse will make 3 strokes on the skin with the palmar side of the fingers of the non-dominant hand at the injection site, simultaneously with the 3rd stroke, the needle will be removed from the baby's skin (Stage 4).
  Arms: Helfer skin tap technique

SUMMARY:
This study will be conducted to determine the effect of mechanical vibration and Helfer Skin Tap technique applied during intramuscular vaccinations on procedural pain level, crying time and procedure time in healthy infants.

DETAILED DESCRIPTION:
Vaccination is one of the painful procedures routinely performed in infants. The pain experienced by the infant negatively affects the prognosis of the disease, the infant's behavior, the harmony with the environment, the development of the brain and senses, as well as the family infant interaction. Nonpharmacologic methods have been found to be effective in alleviating pain during interventions that cause pain caused by medical procedures that infants frequently encounter. Mechanical vibration and Helfer skin tap technique are effective methods that can be used in nonpharmacologic procedural pain management.

Studies have commonly used parent-related methods (kangaroo care, mother/ father cuddling, breastfeeding, etc.) for neonatal pain management during vaccine administrations. In units where access to the parent is not always possible, nonpharmacologic pain methods that can be used independently of the parent can be used in the management of needle related acute pain. In addition, no study was found in the literature comparing the effect of mechanical vibration and Helfer skin tap technique on hepatitis B and DTaP-IPV-Hib vaccinations-related pain. This study will be investigated the effects of mechanical vibration and Helfer skin tap technique methods on procedural pain, crying time and duration of the procedure during intramuscular vaccinations in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy term infants
* born at 38-42 weeks gestational week,
* birth weight 2500-4400 g,
* in stable health,
* able to carry out vital activities without support,
* babies ordered third dose Hepatitis B vaccine by the doctor

Exclusion Criteria:

* with a genetic or congenital anomaly,
* neurological, cardiological and metabolic diseases,
* in need of respiratory support,
* acute or chronic illness that causes pain,
* a complication of childbirth,
* nerve damage or deformity in the extremity to be vaccinated, scar tissue or incision in the vastus lateralis region.

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Procedural pain score: FLACC Pain Scale | 1 min before, during, 1 min after and 3 min after the painful procedure, an average of 4-5 minutes
  The FLACC scale includes the evaluation of five basic behavioural categories. The validity and reliability of the Turkish version of the Pain Diagnostic Scale (FLACC) was conducted. Each of facial expressions, leg movements, activity, crying, and consolability parameters also consists of three sub-items. The items are scored as 0, 1, and 2 point(s) respectively, with total score ranging between 0 to 10 point(s). The "0" point shows that there is no pain, 1-3 points refer to mild pain, 4-6 points refer to moderate pain, and 7-10 points refer to severe pain in infants.

SECONDARY OUTCOMES:
Crying time during the procedure | Through painful procedure completion, an average of 4 minutes
  Total crying time during the procedure is the time the newborn cries between 1 min before and 3 min after the painful procedure.
Length of procedure time | Through painful procedure completion, an average of 60 seconds
  For vaccine administration, it is the time between when the needle is inserted into the skin and when it is removed from the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: September through November of 2025
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Avan Antepli N, Bilsin Kocamaz E, Gungormus Z. The Effect of Vibration on Pain During Heel Lance Procedures in Newborns: A Randomized Controlled Trial. Adv Neonatal Care. 2022 Apr 1;22(2):E43-E47. doi: 10.1097/ANC.0000000000000918. PMID 34334677
- [Background] McGinnis K, Murray E, Cherven B, McCracken C, Travers C. Effect of Vibration on Pain Response to Heel Lance: A Pilot Randomized Control Trial. Adv Neonatal Care. 2016 Dec;16(6):439-448. doi: 10.1097/ANC.0000000000000315. PMID 27533335
- [Background] Baba LR, McGrath JM, Liu J. The efficacy of mechanical vibration analgesia for relief of heel stick pain in neonates: a novel approach. J Perinat Neonatal Nurs. 2010 Jul-Sep;24(3):274-83. doi: 10.1097/JPN.0b013e3181ea7350. PMID 20697246
- [Background] Guven SD, Cakirer Calbayram N. The effect of Helfer skin tap technique on hepatitis B vaccine intramuscular injection pain in neonates: A randomized controlled trial. Explore (NY). 2023 Mar-Apr;19(2):238-242. doi: 10.1016/j.explore.2022.09.001. Epub 2022 Sep 8. PMID 36115789